CLINICAL TRIAL: NCT04263766
Title: The Role of Different Prefrontal Areas in Visual Metacognition
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Georgia Institute of Technology (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: H20033; 5R01MH119189 (NIH)
Record Dates: First submitted 2020-02-07; First posted 2020-02-11 (Actual); Results first posted 2023-09-15 (Actual); Last update posted 2023-09-15 (Actual); Status verified 2023-08

CONDITIONS: Healthy
Keywords: Transcranial Magnetic Stimulation; Metacognition; Prefrontal Cortex
MeSH Terms: interventions — Transcranial Magnetic Stimulation

STUDY DESIGN:
Intervention Model Description: TMS manipulation. Within-subjects design. Each participant will receive TMS to three different sites: DLPFC, aPFC, and a control site.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Healthy Adult Volunteers (Experimental): The experiment has a within-subject design where each subject will receive TMS to different brain areas. The analysis will involve comparing the effects of TMS to different regions.
  Interventions: Other: Transcranial magnetic stimulation

INTERVENTIONS:
Other: Transcranial magnetic stimulation — TMS will be delivered to different brain areas in order to establish their contribution to visual metacognition.

SUMMARY:
The study will use transcranial magnetic stimulation (TMS) to investigate the causal role of different brain regions during visual perception. TMS is a well-established technique used by hundreds of labs in the world. The risks associated with the technique are well understood and can be minimized by strict adherence to established safety guidelines. In the proposed study, the investigators will use TMS to specifically address the topic of how metacognitive evaluation is supported by the two prefrontal areas: the dorsolateral prefrontal cortex (DLPFC) and the anterior prefrontal cortex (aPFC). The data will be collected from healthy adults and will ultimately deepen the investigator's understanding of the mechanisms behind the normal processes related to confidence generation and metacognition.

DETAILED DESCRIPTION:
Participants will complete a task on visual perception and receive TMS in order to assess which regions of the brain are important for confidence generation in perceptual tasks. The task will involve judging the identity of visual stimuli (oriented black-and-white gratings) and providing a confidence rating on the judgment that they performed.

The researchers will deliver TMS to several brain regions such as the anterior prefrontal cortex (aPFC), dorsolateral prefrontal cortex (DLPFC), and a control site. The researchers will then investigate participants' accuracy and confidence levels depending on where TMS was delivered. The researchers expect that aPFC TMS will decrease the metacognitive sensitivity of the participants, whereas DLPFC TMS will decrease their average confidence level. TMS will be delivered time locked to the onset of the stimulus and the researchers will investigate what is the critical period of involvement of a given region.

The TMS protocol is well within the established safety limits. Participants will be required to fill out screening and demographic forms delivered at the Center for Advanced Brain Imaging (CABI). In order to dose appropriately the TMS stimulation, it is necessary to perform motor threshold determination. Motor threshold (MT) is defined as the minimum magnetic flux needed to elicit a visual hand twitch (in the contralateral first dorsal interosseus muscle). MT is the standard in the field for determining the intensity of TMS for each individual to reduce seizure risk. The scalp region producing the largest hand twitch will be identified. At that scalp location, the lowest TMS intensity able to elicit 5 visible twitches in 10 trials at this site will be determined. Individual MT will be used to determine the intensity of stimulation for each individual, as recommended by safety guidelines. This procedure usually takes about 5 minutes and also serves the purpose of acquainting participants to TMS stimulation. In this study, the researchers will use intensities between 100 and 120% of MT, even though the safety guidelines allow for stimulation intensities of at least 130% of MT.

ELIGIBILITY:
Inclusion Criteria:

* right-handed
* adults 18-40
* with normal or corrected-to-normal vision

Exclusion Criteria:

* history of seizures
* family history of epilepsy
* stroke
* severe headaches
* metal anywhere in the head (excluding the mouth)
* cardiac pacemakers
* current use of medication for neurological or psychiatric conditions

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 76 (Actual)
Dates: Start 2022-02-22 (Actual); Primary Completion 2022-08-31 (Actual); Study Completion 2022-08-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dobromir A. Rahnev, Ph.D., Principal Investigator — Georgia Institute of Technology
Locations (1):
- Center for Advance Brain Imaging, Atlanta, Georgia, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- DLPFC Group: The experiment has a within-subject design where each subject will receive TMS to DLPFC at different time point (0 ms, 200 ms, 300 ms, 400 ms, and 500 ms) after the stimulus presentation.
- Vertex Group: The experiment has a within-subject design where each subject will receive TMS to vertex at different time point (0 ms, 200 ms, 300 ms, 400 ms, and 500 ms) after the stimulus presentation.
Period: Overall Study
Arm/Group | DLPFC Group | Vertex Group
Started | 50 | 26
Completed | 43 | 19
Not Completed | 7 | 7
Not completed — Withdrawal by Subject | 6 | 4
Not completed — Lack of Efficacy | 1 | 3

BASELINE CHARACTERISTICS:
Groups:
- DLPFC Group: The experiment has a within-subject design where each subject will receive TMS (Transcranial magnetic stimulation) at DLPFC at different time point (0 ms, 200 ms, 300 ms, 400 ms, 500 ms) after the stimulus presentation in order to reveal the timing of confidence computation in DLPFC.
- Vertex Group: The experiment has a within-subject design where each subject will receive TMS (Transcranial magnetic stimulation) at vertex at different time point (0 ms, 200 ms, 300 ms, 400 ms, 500 ms) after the stimulus presentation in order to reveal the timing of confidence computation in DLPFC.
- Total: Total of all reporting groups
Arm/Group | DLPFC Group | Vertex Group | Total
Number analyzed (Participants) | 50 | 26 | 76
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: Some of the participants didn't provide the date of birth.
  years
    number analyzed (Participants) | 34 | 19 | 53
    (all) | 20.75 (1.81) | 20.96 (10.18) | 20.86 (2.61)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 23 | 12 | 35
  Male | 27 | 14 | 41
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 32 | 16 | 48
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 3 | 1 | 4
  White | 14 | 9 | 23
  More than one race | 1 | 0 | 1
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 50 | 26 | 76

OUTCOME MEASURES:

1. Primary Outcome: Average Confidence Difference With the 0 ms Condition
Description: The average confidence difference for each delay condition and the 0 ms condition for each group (DLPFC or vertex). Confidence was self-reported together with the decision on a 4-point scale with the minimum score being one (not confident at all) and the highest score being four (very confident). The range of the scale is 1 (not confident at all) to 4 (very confident).
Time Frame: 6 months
Population: The analysis population is after the exclusion of subjects who have their 0 ms condition accuracy 3.5% lower than the average accuracy of all delay conditions
Measure: Mean (Standard Deviation); unit: score on a scale (1-4)
Groups:
- DLPFC-200 ms: The study features a within-subject design in which subjects receive TMS at DLPFC at 5 different time points (0 ms, 200 ms, 300 ms, 400 ms, and 500 ms) after stimulus presentation. This arm is for the data of subjects who receive TMS at DLPFC, for 200 ms condition. The measurement is the confidence difference between the 200 ms condition and the 0 ms condition for DLPFC group.
- DLPFC-300 ms: The study features a within-subject design in which subjects receive TMS at DLPFC at 5 different time points (0 ms, 200 ms, 300 ms, 400 ms, and 500 ms) after stimulus presentation. This arm is for the data of subjects who receive TMS at DLPFC, for 200 ms condition. The measurement is the confidence difference between the 300 ms condition and the 0 ms condition for DLPFC group.
- DLPFC-400 ms: The study features a within-subject design in which subjects receive TMS at DLPFC at 5 different time points (0 ms, 200 ms, 300 ms, 400 ms, and 500 ms) after stimulus presentation. This arm is for the data of subjects who receive TMS at DLPFC, for 200 ms condition. The measurement is the confidence difference between the 400 ms condition and the 0 ms condition for DLPFC group.
- DLPFC-500 ms: The study features a within-subject design in which subjects receive TMS at DLPFC at 5 different time points (0 ms, 200 ms, 300 ms, 400 ms, and 500 ms) after stimulus presentation. This arm is for the data of subjects who receive TMS at DLPFC, for 200 ms condition. The measurement is the confidence difference between the 500 ms condition and the 0 ms condition for DLPFC group.
- Vertex-200 ms: The study features a within-subject design in which subjects receive TMS at vertex at 5 different time points (0 ms, 200 ms, 300 ms, 400 ms, and 500 ms) after stimulus presentation. This arm is for the data of subjects who receive TMS at vertex, for 200 ms condition. The measurement is the confidence difference between the 200 ms condition and the 0 ms condition for vertex group.
- Vertex-300 ms: The study features a within-subject design in which subjects receive TMS at vertex at 5 different time points (0 ms, 200 ms, 300 ms, 400 ms, and 500 ms) after stimulus presentation. This arm is for the data of subjects who receive TMS at vertex, for 200 ms condition. The measurement is the confidence difference between the 300 ms condition and the 0 ms condition for vertex group.
- Vertex-400 ms: The study features a within-subject design in which subjects receive TMS at vertex at 5 different time points (0 ms, 200 ms, 300 ms, 400 ms, and 500 ms) after stimulus presentation. This arm is for the data of subjects who receive TMS at vertex, for 200 ms condition. The measurement is the confidence difference between the 400 ms condition and the 0 ms condition for vertex group.
- Vertex-500 ms: The study features a within-subject design in which subjects receive TMS at vertex at 5 different time points (0 ms, 200 ms, 300 ms, 400 ms, and 500 ms) after stimulus presentation. This arm is for the data of subjects who receive TMS at vertex, for 200 ms condition. The measurement is the confidence difference between the 500 ms condition and the 0 ms condition for vertex group.
Arm/Group | DLPFC-200 ms | DLPFC-300 ms | DLPFC-400 ms | DLPFC-500 ms | Vertex-200 ms | Vertex-300 ms | Vertex-400 ms | Vertex-500 ms
Number analyzed (Participants) | 31 | 31 | 31 | 31 | 16 | 16 | 16 | 16
score on a scale (1-4) | 0.14 (0.15) | 0.14 (0.15) | 0.14 (0.14) | 0.15 (0.17) | -0.01 (0.05) | -0.04 (0.08) | -0.04 (0.10) | -0.04 (0.11)
Statistical Analysis 1: Comparison: DLPFC-200 ms vs DLPFC-300 ms vs DLPFC-400 ms vs DLPFC-500 ms vs Vertex-200 ms vs Vertex-300 ms vs Vertex-400 ms vs Vertex-500 ms; Our null hypothesis is TMS to DLPFC would not lead to a significant change in confidence across all 4 delay conditions compared to TMS to the vertex; Test type: Equivalence — We tested whether TMS delivered to DLPFC had a difference effect on confidence compared to delivered to Vertex; p < .001, t-test, 2 sided
Statistical Analysis 2: Comparison: DLPFC-200 ms vs DLPFC-300 ms vs DLPFC-400 ms vs DLPFC-500 ms vs Vertex-200 ms vs Vertex-300 ms; Test type: Equivalence — We tested whether TMS to DLPFC leads to equivalent increase in confidence for four delay conditions; p = 0.99, ANOVA
Statistical Analysis 3: Comparison: Vertex-200 ms vs Vertex-300 ms vs Vertex-400 ms vs Vertex-500 ms; Test type: Equivalence — We tested whether TMS delivered to Vertex leads to a same effect on confidence regardless of the delay conditions; p = 0.83, ANOVA

2. Primary Outcome: Average Mratio Difference With the 0 ms Condition
Description: The average Mratio difference for each delay condition and the 0 ms condition for each group (DLPFC or vertex). The Mratio is derived from signal detection theoretical modeling of the observer's decision and confidence response. It is the ratio of two measures: the observer's metacognitive sensitivity (meta-d', the ability to discriminate between correct and incorrect responses) and the observer's stimulus sensitivity (d', the ability to discriminate between the two stimulus classes). The Mratio could be calculated from subjects' self-rated confidence together with task performance.
Time Frame: 6 month
Population: The analysis population is after the exclusion of subjects whose 0 ms condition accuracy is 3.5% lower than the average accuracy of all four delay conditions.
Measure: Mean (Standard Deviation); unit: Ratio
Groups:
- DLPFC-200 ms: The study features a within-subject design in which subjects receive TMS at DLPFC at 5 different time points (0 ms, 200 ms, 300 ms, 400 ms, and 500 ms) after stimulus presentation. This arm is for the data of subjects who receive TMS at DLPFC, for 200 ms condition. The measurement is the Mratio difference between the 200 ms condition and the 0 ms condition for DLPFC group.
- DLPFC-300 ms: The study features a within-subject design in which subjects receive TMS at DLPFC at 5 different time points (0 ms, 200 ms, 300 ms, 400 ms, and 500 ms) after stimulus presentation. This arm is for the data of subjects who receive TMS at DLPFC, for 200 ms condition. The measurement is the Mratio difference between the 300 ms condition and the 0 ms condition for DLPFC group.
- DLPFC-400 ms: The study features a within-subject design in which subjects receive TMS at DLPFC at 5 different time points (0 ms, 200 ms, 300 ms, 400 ms, and 500 ms) after stimulus presentation. This arm is for the data of subjects who receive TMS at DLPFC, for 200 ms condition. The measurement is the Mratio difference between the 400 ms condition and the 0 ms condition for DLPFC group.
- DLPFC-500 ms: The study features a within-subject design in which subjects receive TMS at DLPFC at 5 different time points (0 ms, 200 ms, 300 ms, 400 ms, and 500 ms) after stimulus presentation. This arm is for the data of subjects who receive TMS at DLPFC, for 200 ms condition. The measurement is the Mratio difference between the 500 ms condition and the 0 ms condition for DLPFC group.
- Vertex-200 ms: The study features a within-subject design in which subjects receive TMS at vertex at 5 different time points (0 ms, 200 ms, 300 ms, 400 ms, and 500 ms) after stimulus presentation. This arm is for the data of subjects who receive TMS at vertex, for 200 ms condition. The measurement is the Mratio difference between the 200 ms condition and the 0 ms condition for vertex group.
- Vertex-300 ms: The study features a within-subject design in which subjects receive TMS at vertex at 5 different time points (0 ms, 200 ms, 300 ms, 400 ms, and 500 ms) after stimulus presentation. This arm is for the data of subjects who receive TMS at vertex, for 200 ms condition. The measurement is the Mratio difference between the 300 ms condition and the 0 ms condition for vertex group.
- Vertex-400 ms: The study features a within-subject design in which subjects receive TMS at vertex at 5 different time points (0 ms, 200 ms, 300 ms, 400 ms, and 500 ms) after stimulus presentation. This arm is for the data of subjects who receive TMS at vertex, for 200 ms condition. The measurement is the Mratio difference between the 400 ms condition and the 0 ms condition for vertex group.
- Vertex-500 ms: The study features a within-subject design in which subjects receive TMS at vertex at 5 different time points (0 ms, 200 ms, 300 ms, 400 ms, and 500 ms) after stimulus presentation. This arm is for the data of subjects who receive TMS at vertex, for 200 ms condition. The measurement is the Mratio difference between the 500 ms condition and the 0 ms condition for vertex group.
Arm/Group | DLPFC-200 ms | DLPFC-300 ms | DLPFC-400 ms | DLPFC-500 ms | Vertex-200 ms | Vertex-300 ms | Vertex-400 ms | Vertex-500 ms
Number analyzed (Participants) | 31 | 31 | 31 | 31 | 16 | 16 | 16 | 16
Ratio | 0.014 (0.959) | 0.087 (0.429) | 0.043 (0.586) | 0.070 (0.467) | -0.211 (0.453) | -0.170 (0.436) | 0.043 (0.386) | 0.077 (0.432)
Statistical Analysis 1: Comparison: DLPFC-200 ms vs DLPFC-300 ms vs DLPFC-400 ms vs DLPFC-500 ms vs Vertex-200 ms vs Vertex-300 ms vs Vertex-400 ms vs Vertex-500 ms; Our null hypothesis is TMS to DLPFC would not lead to a significant change in Mratio across all 4 delay conditions compared to TMS to the vertex; Test type: Equivalence — We used a two-way ANOVA to test whether TMS affected Mratio differently for DLPFC and Vertex and across different delay conditions; p > 0.19, ANOVA

ADVERSE EVENTS:
Time Frame: 6 months
Description: Any event that deviate from regular data collection.
Arm/Group | DLPFC Group | Vertex Group
All-Cause Mortality (participants affected / at risk) | 0/50 | 0/26
Serious Adverse Events (participants affected / at risk) | 0/50 | 0/26
Other Adverse Events (participants affected / at risk) | 0/50 | 0/26

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2023-06-12): https://cdn.clinicaltrials.gov/large-docs/66/NCT04263766/Prot_SAP_001.pdf
  • Informed Consent Form (2021-11-16): https://cdn.clinicaltrials.gov/large-docs/66/NCT04263766/ICF_000.pdf